CLINICAL TRIAL: NCT01233947
Title: A Randomized Phase II Study of AFP464 +/- Faslodex in ER Positive Breast Cancer Patients Who Had Progressed on Aromatase Inhibitor (AI) Therapy
Brief Title: Study of AFP464 +/- Faslodex in ER + Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Tigris Pharmaceuticals (Industry)
Responsible Party: Binh Nguyen, MD PhD / Chief Medical Officer, Tigris Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TG-AFP-003
Record Dates: First submitted 2010-11-01; First posted 2010-11-03 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms | interventions — aminoflavone; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AFP464 (Experimental): 74 mg/m2 AFP464 administered as a 3 hour IV infusion on Days 1 and 8 of a 21-day cycle.
  Interventions: Drug: AFP464
- AFP464 + Faslodex (Experimental): AFP464 administered as a 3 hour IV infusion on Days 1 and 8 of a 21-day cycles and Faslodex administered per package label.
  Interventions: Drug: AFP464 + Faslodex

INTERVENTIONS:
Drug: AFP464 — AFP464 administered as a 3-hour IV infusion on Days 1 and 8 of a 21-day cycle
  Other Names: (aminoflavone)
  Arms: AFP464
Drug: AFP464 + Faslodex — AFP464 administered as a 3-hour IV infusion on Days 1 and 8 of a 21-day cycles and faslodex administered per the package label
  Other Names: (aminoflavone) + (Fulvestrant)
  Arms: AFP464 + Faslodex

SUMMARY:
AFP464 is an investigational agent which may be effective in the treatment of cancer. The purpose of this study is to test the efficacy of AFP464 +/- Faslodex in ER+ breast cancer patients.

DETAILED DESCRIPTION:
This is a randomized, open-label study. Patients will be randomized in a 1:1 ratio to single arm AFP464, or AFP464+Faslodex. Patients will be treated until disease progression is noted.

ELIGIBILITY:
Inclusion Criteria:

* proven breast cancer, ER+ status; progression on an aromatase inhibitor; measurable disease or evaluable disease with serum CA27.29>=50 U/mL; adequate bone marrow, liver and renal function; DLco grade 0 or 1.

Exclusion Criteria:

* HER2 positive, thoracic radiotherapy or symptomatic pulmonary disease, brain metastases,

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-05; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Clinical Benefit Response | 6 months
  Clinical Benefit Response (CBR) defined as Complete Response, Partial Response or Stable Disease for 6 months.

SECONDARY OUTCOMES:
Progression Free Survival | 6 months
  Determination of progression free survival
Number of participants with adverse events | 6 months
  Determination of the number of patients who experience adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Joanne L. Blume, M.D., Principal Investigator — Texas Oncology-Baylor Charles A. Sammons Cancer Center
Locations (1):
- Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas, United States